CLINICAL TRIAL: NCT01087853
Title: The Effects of Balanced and Unbalanced Crystalloids and Colloids on Serum Biochemistry and Visceral Blood Flow: A Two Phase, Double Blind, Randomised Crossover Study
Brief Title: The Effect of Crystalloids and Colloids on Visceral Blood Flow
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Dileep Lobo, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 09063; 2009-014774-18 (EudraCT Number)
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Fluid Overload; Water Electrolyte Imbalance; Acid Base Imbalance
Keywords: Fluid Therapy; Water Electrolyte Imbalance; Acid Base Imbalance; Renal Circulation; Magnetic Resonance Imaging
MeSH Terms: conditions — Edema; Water-Electrolyte Imbalance; Acid-Base Imbalance | interventions — Crystalloid Solutions; Colloids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase A1: Plasmalyte (Active Comparator): Plasmalyte
  Interventions: Drug: Crystalloid
- Phase A2: 0.9% Saline (Active Comparator): 0.9% Saline
  Interventions: Drug: Crystalloid
- Phase B1: PlasmaVolume (Active Comparator): PlasmaVolume
  Interventions: Drug: Colloid
- Phase B2: Voluven (Active Comparator): Voluven
  Interventions: Drug: Colloid

INTERVENTIONS:
Drug: Crystalloid — 2 litres intravenous infusion in 60 minutes
  Arms: Phase A1: Plasmalyte; Phase A2: 0.9% Saline
Drug: Colloid — 1 litre intravenous infusion over 30 minutes
  Arms: Phase B1: PlasmaVolume; Phase B2: Voluven

SUMMARY:
Patients often require fluid replacement during and after an operation. This is usually given through veins in the arm using an intravenous cannula and doctors have traditionally used fluid containing sodium chloride (saline). However accumulating evidence suggests that large infusions of saline are associated with adverse physiological effects including acidification of the blood and a rise in potassium and chloride levels. Studies in animals have shown that high levels of chloride in the blood and excess saline can cause blood vessels in the kidney to constrict leading possibly to a decrease in kidney function. Improvement in acid-base balance and kidney function may be observed with balanced solutions containing constituents that are more closely matched to the body's own fluid composition. However, little is known about the physiological effects of these solutions as they have only recently been developed.

Magnetic resonance imaging (MRI) is a radiological modality which can now assess blood flow and supply of the kidney noninvasively without the need for the injection of radiological dyes known as contrast agents. This is now of major importance due to the possible adverse effects of MRI contrast agents leading to Nephrogenic Systemic Fibrosis (NSF), a progressive disease which has been observed in some kidney patients after receiving 'gadolinium based' contrast agents. This has therefore led to increased interest and demand for noncontrast based imaging methods. In this study we aim to compare the effects of balanced versus unbalanced fluid infusions in healthy human volunteers:

We will aim to measure:

1. Blood biochemical composition and acidity
2. Kidney function and supply as measured by dynamic MRI

DETAILED DESCRIPTION:
Type of Study: Two phase double blind, randomised crossover study. In phase A (crystalloid), we will compare the effects of Plasmalyte 148 with 0.9% saline and in phase B (colloid) we will compare the effects of PVR with Voluven.

Participants will either be involved in phase A or phase B not both. In each phase participants will receive a randomly assigned fluid and then the comparator fluid 1 week later.

Subject selection: 24 healthy, male volunteers, (12 for each phase) between the age of 18 and 40, and weighing between 65 and 80 kg will be recruited for of the study. Informed consent will be obtained before entering volunteers into the study.

Study Protocol: Volunteers will report for the study at 09.00 hours after a fast from midnight and having abstained from alcohol, nicotine, tea and coffee for at least 24 hours. After voiding of the bladder, height will recorded to the nearest 0.01 m, weight measured to the nearest 0.1 kg using Avery 3306ABV scales (Avery Berkel, Royston, UK), and body mass index calculated.

Any urine passed over a 24 hour period from the start of the infusion will be collected for measurement of creatinine clearance, osmolality and electrolytes. Two venous cannulae will be inserted, one in each forearm and blood will be sampled for full blood count, haemoglobin, electrolytes, creatinine, albumin and osmolality. A venous blood gas sample will also be obtained to calculate base excess. Serum and urinary osmolality will be measured on a Fiske 2400 Osmometer (Vitech Scientific Ltd., Partridge Green, West Sussex, UK) using a freezing point depression method which has a coefficient of variance (CV) of 1.2%. A Vitros 950 analyser (Ortho Clinical Diagnostics, Amersham, UK) will be used to measure serum sodium (CV 0.6%), potassium (CV 1.0%), magnesium, chloride (CV 1.1%), bicarbonate, (CV 4.0%), urea (CV 2.0%) and albumin (CV 1.6%). Strong ion difference will be calculated by subtracting the serum chloride concentration from the sum of the serum concentrations of sodium and potassium.28 Urinary sodium (CV 1.5%) and potassium (CV 1.5%) will be assayed on a Vitros 250 analyser (Ortho Clinical Diagnostics, Amersham, UK). Haematological parameters will be measured on a Sysmex SE 9500 Analyser (Sysmex UK Ltd., Milton Keynes, UK) using direct current hydrodynamic focusing and cumulative pulse height detection. The CV for haemoglobin and packed cell volume estimation is 11.5%.

In Phase A, 12 subjects will receive 2 litres of 0.9% saline BP (Baxter Health Care, Thetford, UK) or Plasmalyte® (Baxter Health Care, Thetford, UK). The assignment of the initial infused solution will be random followed by the alternate solution at crossover. The crystalloid solution will be infused in the supine position over 60 minutes.

In Phase B, 12 subjects will receive 1 litre of PlasmaVolume® (Baxter Health Care, Thetford, UK) or Voluven® (Fresenius Kabi, Bad Homburg, Germany). The initial infused solution will be randomly assigned and the subject will receive the alternate solution at the crossover timepoint. The starch solution will be infused in the supine position over 30 minutes. A nurse who will not be involved in the study will mask all labels and administration sets on the infusion bags with opaque tape and also perform the randomisation. Randomisation will performed using sequentially numbered paired sealed opaque envelopes. The aforementioned blood tests will be repeated at 30/60 minute intervals for 4 hours. Subjects will be encouraged to void urine as the need arises, and on completion of the study. In addition to laboratory data, time to first void and void volume will be recorded. Postinfusion urine will be pooled and analysed for osmolality, pH and concentrations of electrolytes and NGAL. The crossover experiment will be repeated with the alternate infusion not used in the first study, 7-10 days later. Participation in the crossover phase will be postponed one week if the baseline laboratory work shows continued effect of hemodilution or phlebotomy with a hematocrit decrease of 3% or greater from the first infusion baseline.

Monitoring of volunteers: Pulse oximetry will be performed continuously during the infusion. Blood pressure will be measured every 15 min for the first two hours and then every 30 min until the end of the study. Infusions will be stopped if there is any evidence of hypersensitivity or anaphylactic reactions or for the following:

The pulse rate rises above 110/minute or falls below 50/minute. The SaO2 falls below 92% The blood pressure rises above 140 mm Hg systolic or 95 mm Hg diastolic The blood pressure falls below 90 mm Hg systolic or 55 mm Hg diastolic The volunteer expresses the desire to have the infusion stopped.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male
* Aged between 18 and 40 years
* Weight between 65 and 80 kilograms
* Able to give informed consent

Exclusion Criteria:

* Chronic medical conditions
* Use of any regular medications
* History of substance abuse
* Known hypersensitivity to study infusion fluids
* Contraindications to MRI scanning

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary end point of each phase of this study will be a 6 mmol difference in serum chloride concentration after infusion of the balanced and unbalanced crystalloids and colloids. | Phase A: Times 0, 60, 90, 120, 180 and 240 min and Phase B: Times 0, 30, 60, 120, 180 and 240 min

SECONDARY OUTCOMES:
Changes in blood volume, renal and superior mesenteric arterial blood flow and vessel diameter. | Phase A: Times 0, 60, 90, 120, 180 and 240 min and Phase B: Times 0, 30, 60, 120, 180 and 240 min

CONTACTS AND LOCATIONS:
Overall Officials: Dileep Lobo, MBBS MD FRCS, Principal Investigator — University of Nottingham
Locations (1):
- Brain and Body MRI Centre, University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Derived] Chowdhury AH, Cox EF, Francis ST, Lobo DN. A randomized, controlled, double-blind crossover study on the effects of 2-L infusions of 0.9% saline and plasma-lyte(R) 148 on renal blood flow velocity and renal cortical tissue perfusion in healthy volunteers. Ann Surg. 2012 Jul;256(1):18-24. doi: 10.1097/SLA.0b013e318256be72. PMID 22580944